CLINICAL TRIAL: NCT06557889
Title: Reduction in the Number of Chemotherapy Cycles in Combination With Pembrolizumab in First-line Treatment of PD-L1-positive Recurrent or Metastatic Head and Neck Squamous Cell Carcinomas
Acronym: REDUCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24VADS04
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Squamous Cell Carcinoma of Head and Neck; Pembrolizumab; Cisplatin; Carboplatin; 5-fluorouracil
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with PD-L1-positive recurrent or metastatic squamous cell carcinoma of the head and neck (Experimental)
  Interventions: Drug: Pembrolizumab + Cisplatin/Carboplatin + 5-FU

INTERVENTIONS:
Drug: Pembrolizumab + Cisplatin/Carboplatin + 5-FU — * 4 cycles of combination treatment: 4 cycles of pembrolizumab (200 mg IV on Day 1 of each 3-week cycle) in combination with chemotherapy with platinum salts (cisplatin (100 mg/m2 IV on Day 1 of each 3-week cycle) or carboplatin (AUC 5 IV on Day 1 of each 3-week cycle), at the investigator's choice) and 5-FU (1000 mg/m2/day IV continuous from Day 1-4 of each 3-week cycle).
  * Maintenance phase: pembrolizumab is continued as monotherapy for up to 24 months of treatment in total (from the first injection of cycle 1).

SUMMARY:
This is a phase II, prospective, non-randomized, single-arm, multicentric study to evaluate the activity and safety of treatment with 4 cycles (instead of 6) of chemotherapy (platinum (cisplatin or carboplatin) and 5-Fluorouracil) in combination with pembrolizumab for the first-line treatment of CPS PD-L1 positive recurrent or metastatic head and neck squamous cell carcinoma.

A total of 86 patients will have to be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old on the day of signing the informed consent.
2. Diagnosis of histologically proven recurrent or metastatic squamous cell carcinoma of the head and neck not accessible to treatment with curative intent.
3. Patients must not have received previous systemic therapy administered in the context of recurrent or metastatic disease.
4. If the patient received chemotherapy with a platinum salt as part of multimodal treatment for locally advanced disease, it must have ended at least 6 months before signing the consent.
5. Eligible primary tumor locations are the oropharynx, oral cavity, hypopharynx and larynx. Subjects cannot have a primary tumor site (any histology) in the nasopharynx, sinuses, nasal cavity, salivary glands, or skin.
6. Documented Combined Positive Score (CPS) PD-L1 ≥ 1 (determined according to local practices in each center) Note: the CPS score can be performed on a new biopsy or on an archived tumor specimen, without date limitation.
7. Have measurable disease on CT-scan (or on MRI of the neck if it provides a better measurement of the primary tumor according to standard practice and the investigator judgement) according to RECIST 1.1 as determined by the investigator. Tumor lesions located in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Note : In case of neck MRI assessment, the chest, abdominal, and pelvic CT scan must be performed in addition to assess potential metastases.
8. Have a performance status of 0 or 1 on the ECOG performance scale.
9. Demonstrate adequate organ function as defined in the protocol.
10. Have HPV status test results for oropharyngeal cancers defined as a p16 immunohistochemical (IHC) test (determined according to local practices in each center).

    Note: Cancers of the oral cavity, hypopharynx, and larynx are not required to perform HPV testing by p16 IHC because, by convention, these tumor locations are assumed to be HPV negative.
11. Female subjects of childbearing potential must have a negative pregnancy test within 72 hours prior to receiving the first dose of study treatment.
12. Female subjects of childbearing potential must be willing to follow at least one method of contraception or be surgically sterile, or abstain from heterosexual activity for the duration of the study and until 4 months for pembrolizumab, 6 months for carboplatin and 5-fluorouracil, and 7,5 months for cisplatin after the last dose of study treatment respectively for each molecule. Subjects of childbearing potential are those who have not been surgically sterilized and who had menstruation in the last 12 months.

    Note: Abstinence is acceptable if it is the subject's usual lifestyle and preferred method of contraception.
13. Male subjects must agree to use at least one method of contraception for the duration of the study and until 180 days after the last dose of study treatment.

    Note: Abstinence is acceptable if it is the subject's usual lifestyle and preferred method of contraception.
14. Signed written informed consent
15. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol
16. Patient affiliated to a Social Health Insurance in France

Exclusion Criteria:

1. Has a disease accessible to local treatment with curative intent.
2. Has a progressive disease within six months following the end of primary treatment with curative intent, if this treatment included systemic treatment with platinum salt.
3. Has a complete DPD enzyme deficiency, suggested by an uracilemia > or equal to 150 ng/mL.
4. Has a contraindication to full dose use of a platinum salt, 5-Fluorouracil, or pembrolizumab, in the opinion of the investigator (dose reductions in cycle 1 are not authorized, except in the case of adaptation of the 5-FU due to partial DPD deficiency); the investigator must refer to the SmPC of the products used in this trial (carboplatin, cisplatin, 5-fluorouracil, and pembrolizumab).
5. The patient must not have received antibiotics within 14 days before inclusion in the trial.
6. Received radiotherapy (or other non-systemic therapy) within 2 weeks prior to inclusion.
7. Subject has not fully recovered (i.e. ≤ Grade 1) from adverse events due to previously administered treatment.

   Note: Subjects with neuropathy ≤ Grade 2, alopecia ≤ Grade 2, or laboratory values not exceeding the limits in Table 1 (See the protocol) are an exception to this criterion and may be eligible for the study Note: If the subject has undergone major surgery, they must have adequately recovered from the toxicity and/or complications of the procedure before starting treatment.
8. Currently participating in and receiving study treatment, or has participated in a study of an investigational agent, or used an investigational device, within 4 weeks prior to the first dose of treatment.

   Note: Participation in the follow-up phase of a previous study is permitted (if the patient is no longer receiving treatment in that study).
9. Has a life expectancy of less than 3 months and/or has a rapidly progressing illness (eg, tumor bleeding, uncontrolled tumor pain) in the opinion of the investigator.
10. Has a diagnosis of immunodeficiency or is receiving systemic corticosteroid therapy > 10 mg/day of prednisone equivalent or any other form of immunosuppressive therapy within 7 days before the first dose of trial treatment. The use of corticosteroids as premedication for allergic reactions (e.g., IV contrast) or as prophylactic management of adverse events related to protocol-specified chemotherapies is permitted.
11. Has a diagnosis of a second cancer diagnosed and/or treated within 5 years preceding inclusion, with the exception of: curatively resected basal cell carcinoma of the skin, curatively resected squamous cell carcinoma of the skin, curatively resected in situ cervical cancer and curatively resected in situ breast cancer.

    Note: The 5 year period does not apply to the cancer for which the subject is enrolled in the trial.
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

    Note: Subjects with previously treated brain metastases may participate provided they have been stable (without evidence of progression by imaging using the same imaging modality for each assessment, either MRI or CT) for at least 4 weeks prior to the first dose of trial treatment, and without neurological symptoms, have no signs of new or progressing brain metastases, and are not using steroids > 10mg/day of prednisone equivalent for at least 7 days before study inclusion. This exception does not include carcinomatous meningitis which is excluded regardless of the clinical situation.
13. Active autoimmune disease that has required systemic treatment within the past 2 years (i.e. with the use of corticosteroids or immunosuppressive drugs). Replacement therapy (for example: thyroxine, insulin or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Has undergone solid tissue/organ allograft or hematopoietic allograft.
15. Has a history of or has non-infectious pneumonia requiring corticosteroids.
16. Has an active infection requiring systemic anti-infectious treatment.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that could interfere with the results of the trial or with the subject's participation throughout the duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the investigator.
18. Is pregnant or breastfeeding, or expects to conceive or father children during the planned duration of the trial, beginning the screening visit through and until 4 months for pembrolizumab, 6 months for carboplatin and 5-fluorouracil, and 7,5 months for cisplatin after the last dose of study treatment respectively for each molecule.
19. Has previously received treatment with an anti-PD-1 or anti-PD-L1 agent for the treatment of the cancer for which the patient is included in the trial, whether as part of the primary treatment or as part of the relapse.
20. Has a known history of human immunodeficiency virus (HIV) infection.
21. Has known active hepatitis B or C.
22. Received a live vaccine within 30 days before the planned start of study treatment.
23. Has a known history of hypersensitivity to fluorouracil, carboplatin, cisplatin or pembrolizumab or to any of their excipients, according to the SmPCs of these products.
24. For patient receiving the treatment with 5-fluorouracil: has clinically significant active heart disease or myocardial infarction within 6 months; has received a recent or has a concomitant treatment with brivudine (4 weeks before or after 5-FU).
25. For patient receiving the treatment with cisplatin: has a neuropathy caused by cisplatin, has a hearing problem, has a treatment with phenytoin with prophylactic aim.
26. For patient receiving the treatment with pembrolizumab: has a history of uncontrolled or symptomatic cardiac disease.
27. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
28. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
The endpoint for the activity is defined by the objective response (i.e. complete or partial response) according to the RECIST v1.1 criteria, assessed by the investigator. | 48 months for each patient
  The objective response rate is defined as the ratio of the number of patients with an objective response to the total number of patients.
The endpoint for the safety is defined as the rate of patients with AE leading to all treatment discontinuation. | 24 months for each patient
  This rate is defined as the ratio of the number of patients with AE leading to all treatment discontinuation to the total number of patients.

SECONDARY OUTCOMES:
The objective response rate at 6 months is defined by the presence of an objective response (i.e. complete or partial response) at 6 months according to the RECIST v1.1 criteria, assessed by the investigator. | 6 months for each patient
  It is defined by the ratio of the number of patients presenting an objective response at 6 months to the total number of patients.
Progression-free survival is defined by the time between the date of inclusion and the date on which a first tumor confirmed progression is documented (according to RECIST v1.1 criteria, (Eisenhauer, 2009)) or death from any causes. | 48 months for each patient
  Patients alive and progression free on the date of last news will be censored on the date of last tumor assessment.
Overall survival is defined by the time between the date of inclusion and the date of death from any cause or the date of the last news (Censored Data). | 48 months for each patient
Duration of response is defined in the population of patients with an objective response. | 48 months for each patient
  It is defined by the time between the date of confirmed objective response and the date on which a first confirmed tumor progression is documented (according to RECIST v1.1 criteria, Eisenhauer, 2009) or death from all causes. Patients alive and progression free at last news will be censored on the date of last tumor assessment.
Safety will be assessed according to the toxicity grading of NCI CTCAE v 5.0. | 48 months for each patient

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU Amiens, Amiens
  - Institut Sainte Catherine, Avignon
  - Chu Bordeaux - Hopital Saint André, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Chu Limoges, Limoges
  - Centre Hospitalier Regional de Marseille, Marseille
  - CHU de Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - Chu de Nimes, Nîmes
  - CHU Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - Clinique Pasteur, Toulouse
  - IUCT-O, Toulouse